CLINICAL TRIAL: NCT03785405
Title: A Multicenter Study to Evaluate Long-term Safety and Tolerability of Open Label Sacubitril/Valsartan in Pediatric Patients With Heart Failure Due to Systemic Left Ventricle Systolic Dysfunction Who Have Completed Study CLCZ696B2319
Brief Title: Open-label Extension Study to Evaluate Long-term Safety of Sacubitril/Valsartan in Pediatric Patients With HF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCZ696B2319E1
Record Dates: First submitted 2018-12-20; First posted 2018-12-24 (Actual); Results first posted 2024-07-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Heart Failure
Keywords: heart failure; pediatric; LCZ696; sacubitril/valsartan; open-label study; angiotensin receptor neprilysin inhibitor; PANORAMA-HF
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sacubitril/valsartan (Experimental): single arm, open label sacubitril/valsartan
  Interventions: Drug: sacubitril/valsartan

INTERVENTIONS:
Drug: sacubitril/valsartan — Target dose 3.1 mg/kg bid
  Formulations:
  Tablets (50, 100, 200 mg) Granules [12.5 mg (4 granules), 31.25 mg (10 granules), in capsules] Liquid (1 mg/ml, 4 mg/ml, prepared from tablets)
  Other Names: LCZ696

SUMMARY:
The purpose of this study was to evaluate long-term safety and tolerability and to provide post-trial access to sacubitril/valsartan to eligible participants who successfully completed CLCZ696B2319 (PANORAMA-HF) core study Part 2 as per protocol.

DETAILED DESCRIPTION:
This was a multicenter, open-label long-term extension study for participants who successfully completed PANORAMA-HF core study Part 2 of the trial or who discontinued study drug treatment early in Part 2 due to the implementation of Urgent safety measure (USM) of PANORAMA-HF core study. Provided that they fulfilled the protocol requirements, these patients were eligible to participate in the OLE. Depending on when and where the participant was enrolled, the duration of the study was of a minimum of 1 year, or until receipt of local marketing authorization and commercial availability, or reaching the maximum limit allowed by local regulations, or until Dec-2023, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* On study drug at PANORAMA-HF Part 2 EOS visit. Does not have any significant safety issue

Exclusion Criteria:

* Subject only participated in PANORAMA-HF Part 1 or was a SF in PANORAMA-HF or permanently discontinued study drug in PANORMA-HF Part 2
* Use of investigational drugs within 5 half-lives of enrollment or within 30 days (longer duration); with the exception of PANORAMA-HF study drug (requires >/=36-hour washout before baseline visit)
* History of hypersensitivity or allergy to study treatment, its excipients or drugs of similar chemical class, ACEIs, ARBs, or NEP inhibitor and known/suspected contraindications to sacubitril/valsartan
* Renal vascular hypertension (including renal artery stenosis)
* Significant renal estimated glomerular filtration rate disorder (eGFR calculated using modified Schwartz formula <30% mean GFR for age); hepatic disorder (serum aspartate aminotransferase or alanine aminotransferase > 3 times upper limit of normal); gastrointestinal disorder or biliary disorder
* History of angioedema
* Parents or legal guardians of subject who do not give consent or allow the child to give assent, or inability of patient or parents/legal guardians to follow instructions or comply with follow-up procedures
* Any medical condition(s) that may put the patient at risk in the investigator's opinion or that the investigator deems unsuitable for the study
* Other protocol defined inclusion/exclusion criteria may apply

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 216 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (75):
- United States (15):
  - Novartis Investigative Site, Loma Linda, California
  - Novartis Investigative Site, Los Angeles, California
  - Novartis Investigative Site, Palo Alto, California
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
- Novartis Investigative Site, Salta, Salta Province, Argentina
- Novartis Investigative Site, Innsbruck, Austria
- Novartis Investigative Site, Sofia, Bulgaria
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Toronto, Ontario
- Novartis Investigative Site, Zagreb, Croatia
- Novartis Investigative Site, Prague, Czechia
- Novartis Investigative Site, Helsinki, Finland
- Novartis Investigative Site, Paris, France
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Heidelberg
  - Novartis Investigative Site, Stuttgart
- Novartis Investigative Site, Budapest, Hungary
- India (4):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Kochi, Kerala
  - Novartis Investigative Site, New Delhi, National Capital Territory of Delhi
  - Novartis Investigative Site, New Delhi
- Novartis Investigative Site, Beersheba, Israel
- Italy (7):
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Napoli
- Japan (8):
  - Novartis Investigative Site, Ōbu, Aichi-ken
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Saitama
- Lebanon (2):
  - Novartis Investigative Site, Beirut
  - Novartis Investigative Site, El Achrafiyé
- Poland (2):
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (3):
  - Novartis Investigative Site, Carnaxide, Lisbon District
  - Novartis Investigative Site, Coimbra
  - Novartis Investigative Site, Lisbon
- Russia (2):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Soweto, Gauteng, South Africa
- South Korea (2):
  - Novartis Investigative Site, Yangsan, Gyeongsangnam-do
  - Novartis Investigative Site, Seoul
- Spain (4):
  - Novartis Investigative Site, Córdoba, Andalusia
  - Novartis Investigative Site, Esplugues de Llobregat, Barcelona
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Novartis Investigative Site, Lausanne, Switzerland
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Thailand (2):
  - Novartis Investigative Site, Bangkoknoi, Bangkok
  - Novartis Investigative Site, Bangkok
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir
  - Novartis Investigative Site, Konak-Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2355

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 79 centers in 27 countries: Korea, Republic of(4), United States(15), Bulgaria(1), Italy(7), Thailand(2), Poland(2), Japan(8), Singapore(2), Israel(1), Turkey(3), Taiwan(2), South Africa(1), Portugal(3), Lebanon(2), Canada(2), Switzerland(1), Czech Republic(1), Croatia(1), Argentina(1), Hungary(1), India(4), Germany(5), France(1), Austria(1), Spain(5), Russia(2), Finland(1)
Pre-assignment Details: A 36-hour washout after the last dose of study medication taken in the PANORAMA-HF core study (Visit 416) was required for all participants before starting Open Label Extension study medication.
Groups:
- Age Group 1: Patients 6 years and older receiving open label sacubitril/valsartan 3.1 mg/kg bid
- Age Group 2: Patients 1 year to < 6 years receiving open label sacubitril/valsartan 3.1 mg/kg bid
Period: Overall Study
Arm/Group | Age Group 1 | Age Group 2
Started | 130 | 86
Safety Set (SAF) (All screened participants who received at least one dose of open-label study treatment.) | 130 | 85
Completed | 92 | 74
Not Completed | 38 | 12
Not completed — Adverse Event | 16 | 1
Not completed — Death | 6 | 4
Not completed — Guardian decision | 4 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 8 | 5
Not completed — Participant decision | 2 | 0
Not completed — Other | 1 | 0
Not completed — No treatment was received | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline Participants are based on the Safety Set (SAF) population, as primary analysis are based on the SAF.
Groups:
- Total: Total of all reporting groups
Arm/Group | Age Group 1 | Age Group 2 | Total
Number analyzed (Participants) | 130 | 85 | 215
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.83 (3.864) | 2.94 (1.149) | 8.92 (5.747)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 49 | 109
  Male | 70 | 36 | 106
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  White | 78 | 41 | 119
  Asian | 24 | 23 | 47
  Black or African American | 19 | 10 | 29
  Multiple | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Unknown | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants with at least one Adverse Events (AEs)
Time Frame: to end of study, up to 4,5 years
Population: Safety Set (SAF): All participants who received at least one dose of open-label study treatment during the extension open-label study.
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 1 | Age Group 2
Number analyzed (Participants) | 130 | 85
Participants | 111 | 78

2. Primary Outcome: Number of Participants With Serious Adverse Events
Description: Number of participants with at least one Serious Adverse Events (SAEs)
Time Frame: to end of study, up to 4.5 years
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Age Group 1 | Age Group 2
Number analyzed (Participants) | 130 | 85
Participants | 59 | 25

3. Primary Outcome: Duration of Drug Exposure
Description: Median duration of exposure to sacubitril/valsartan (including temporary interruptions)
Time Frame: Up to 4.5 years
Population: as for outcome 1
Measure: Median (Full Range); unit: Days
Arm/Group | Age Group 1 | Age Group 2
Number analyzed (Participants) | 130 | 85
Days | 894 [23 to 1612] | 951 [62 to 1570]

ADVERSE EVENTS:
Time Frame: Adverse events were reported from first dose of study treatment until end of study treatment plus 30 days post treatment, up to a maximum duration of 4.5 years
Description: Adverse Events are assessed in the safety population.
Groups:
- Total: Total
Arm/Group | Age Group 1 | Age Group 2 | Total
All-Cause Mortality (participants affected / at risk) | 7/130 | 4/85 | 11/215
Serious Adverse Events (participants affected / at risk) | 59/130 | 25/85 | 84/215
Other Adverse Events (participants affected / at risk) | 90/130 | 60/85 | 150/215
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Age Group 1 (N=130) | Age Group 2 (N=85) | Total (N=215)
Splenic cyst (Blood and lymphatic system disorders) | 1 | 0 | 1
Arrhythmia (Cardiac disorders) | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 2
Atrial flutter (Cardiac disorders) | 2 | 0 | 2
Cardiac arrest (Cardiac disorders) | 1 | 0 | 1
Cardiac failure (Cardiac disorders) | 15 | 3 | 18
Cardiac failure acute (Cardiac disorders) | 2 | 2 | 4
Cardiac failure chronic (Cardiac disorders) | 4 | 2 | 6
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1
Dilated cardiomyopathy (Cardiac disorders) | 5 | 0 | 5
Left ventricular dysfunction (Cardiac disorders) | 2 | 0 | 2
Mitral valve incompetence (Cardiac disorders) | 1 | 0 | 1
Pericardial effusion (Cardiac disorders) | 2 | 0 | 2
Pulmonary valve stenosis (Cardiac disorders) | 1 | 0 | 1
Tachycardia induced cardiomyopathy (Cardiac disorders) | 0 | 1 | 1
Torsade de pointes (Cardiac disorders) | 1 | 0 | 1
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 1
Ventricular dysfunction (Cardiac disorders) | 0 | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 2 | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 2 | 1 | 3
Congenital epiblepharon (Congenital, familial and genetic disorders) | 1 | 0 | 1
Cryptorchism (Congenital, familial and genetic disorders) | 1 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1
Abdominal wall haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0 | 1
Dental caries (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 3 | 2 | 5
Chest pain (General disorders) | 5 | 0 | 5
Complication associated with device (General disorders) | 1 | 1 | 2
Medical device site extravasation (General disorders) | 0 | 1 | 1
Medical device site pain (General disorders) | 0 | 1 | 1
Pyrexia (General disorders) | 3 | 3 | 6
Hepatitis (Hepatobiliary disorders) | 1 | 1 | 2
Heart transplant rejection (Immune system disorders) | 1 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 1
COVID-19 (Infections and infestations) | 4 | 4 | 8
COVID-19 pneumonia (Infections and infestations) | 2 | 0 | 2
Cytomegalovirus infection (Infections and infestations) | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 4 | 2 | 6
Gastroenteritis norovirus (Infections and infestations) | 0 | 1 | 1
Influenza (Infections and infestations) | 1 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 2 | 2
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1 | 1
Neutropenic infection (Infections and infestations) | 0 | 1 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 1
Pneumonia (Infections and infestations) | 5 | 4 | 9
Pneumonia aspiration (Infections and infestations) | 1 | 1 | 2
Pneumonia mycoplasmal (Infections and infestations) | 1 | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1 | 1
Pneumonia viral (Infections and infestations) | 0 | 1 | 1
Post procedural infection (Infections and infestations) | 0 | 1 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1 | 1
Pseudomonas infection (Infections and infestations) | 1 | 0 | 1
Respiratory syncytial virus infection (Infections and infestations) | 1 | 1 | 2
Respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Vascular device infection (Infections and infestations) | 0 | 1 | 1
Viral infection (Infections and infestations) | 0 | 1 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1
Ejection fraction decreased (Investigations) | 1 | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0 | 1
Respiratory syncytial virus test positive (Investigations) | 0 | 1 | 1
Staphylococcus test positive (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 2
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Intervertebral disc space narrowing (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1 | 1
Febrile convulsion (Nervous system disorders) | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 1
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0 | 1
Status epilepticus (Nervous system disorders) | 1 | 0 | 1
Device malfunction (Product Issues) | 1 | 0 | 1
Device power source issue (Product Issues) | 1 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 0 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 1
Prerenal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Hypotension (Vascular disorders) | 3 | 1 | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Age Group 1 (N=130) | Age Group 2 (N=85) | Total (N=215)
Abdominal pain (Gastrointestinal disorders) | 10 | 3 | 13
Diarrhoea (Gastrointestinal disorders) | 9 | 9 | 18
Nausea (Gastrointestinal disorders) | 9 | 1 | 10
Vomiting (Gastrointestinal disorders) | 15 | 12 | 27
Chest pain (General disorders) | 8 | 2 | 10
Pyrexia (General disorders) | 15 | 22 | 37
COVID-19 (Infections and infestations) | 23 | 24 | 47
Conjunctivitis (Infections and infestations) | 3 | 5 | 8
Gastroenteritis (Infections and infestations) | 7 | 7 | 14
Influenza (Infections and infestations) | 6 | 8 | 14
Nasopharyngitis (Infections and infestations) | 12 | 14 | 26
Pharyngitis (Infections and infestations) | 6 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 8 | 22 | 30
SARS-CoV-2 test positive (Investigations) | 13 | 1 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 2 | 10
Dizziness (Nervous system disorders) | 14 | 0 | 14
Headache (Nervous system disorders) | 15 | 3 | 18
Cough (Respiratory, thoracic and mediastinal disorders) | 20 | 19 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 0 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 2 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 6 | 6 | 12
Hypotension (Vascular disorders) | 18 | 3 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/05/NCT03785405/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/05/NCT03785405/SAP_001.pdf